CLINICAL TRIAL: NCT00003787
Title: Dietary Intervention in Women Who Have Been Treated For Stage I, Stage II, or Stage III Breast Cancer: Women's Healthy Eating and Living (WHEL) Study
Brief Title: Women's Healthy Eating and Living Study
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, John P. Pierce, Professor, University of California, San Diego
Other Study IDs: UCSD-980919; CDR0000066920 (Registry Identifier: PDQ (Physician Data Query)); UCSD-WHEL; NCI-G99-1508
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, RBC, DNA at five time periods
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention: high fiber, high vegetable, low-fat diet
  Interventions: Behavioral: educational/counseling intervention; Behavioral: therapeutic dietary intervention
- Control: NCI-recommended diet
  Interventions: Behavioral: therapeutic dietary intervention

INTERVENTIONS:
Behavioral: educational/counseling intervention
  Groups: Intervention
Behavioral: therapeutic dietary intervention

SUMMARY:
RATIONALE: Dietary fats, fruits, vegetables, and fiber may affect the risk of breast cancer recurrence.

PURPOSE: Randomized clinical trial to determine the effectiveness of a diet rich in vegetables, fruit, and fiber and low in fat in women who have been treated for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a diet rich in vegetables, fruit, and fiber and low in fat is associated with a longer breast cancer event-free interval in breast cancer survivors. II. Motivate an intervention group of breast cancer survivors to adopt and maintain a dietary pattern that is rich in vegetables, fruit, and fiber and low in fat. III. Demonstrate that the intervention can produce significant changes in circulating carotenoid and estrogen biomarkers compared to a healthy control diet. IV. Test whether the probability of a secondary cancer event is associated with change in self-reported dietary intake, circulating carotenoid concentrations, and circulating estrogen concentrations.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 55 vs 55 and over at time of diagnosis), stage of tumor (stage I and at least 1 cm vs stage II/IIIA), and clinical site. Patients are randomized to one of two healthy dietary regimens: Arm I: Patients are taught to follow a dietary pattern that will produce significant changes in circulating carotenoid and estrogen biomarkers. Arm II: Patients are assigned to follow dietary guidelines established by the National Cancer Institute and the USDA. All patients participate in 24 hour dietary recalls, cooking classes, as well as complete several questionnaires, at baseline and then at 12, 24 or 36, 48, and 72 months; a randomly selected 50% sample participate in recall at 6 months. Patients are followed by telephone every 6 months for an average of 6 years.

PROJECTED ACCRUAL: A total of 3,000 women will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary operable stage I (tumors at least 1 cm), stage II, and stage IIIA invasive breast carcinoma Treatment within the past 4 years by total mastectomy and axillary dissection, or breast sparing surgical removal of cancer with clear macroscopic margins and axillary dissection followed by adjuvant breast radiation No evidence of recurrent disease or new breast cancer since completion of initial local treatment confirmed within the past 6 months by physician evaluation, except stage I mastectomy, for which physician evaluation can be within 1 year prior to randomization Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 70 at time of diagnosis Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: At least 10 years (excluding breast cancer) Hematopoietic: Not specified Hepatic: No cirrhosis Renal: Not specified Other: Not pregnant Accessible geographically and by telephone Able to communicate dietary data via 24-hour food recall Able to commit to the intervention schedule No comorbidity requiring a specific diet or taking a medication which contraindicates consuming a high fiber diet (e.g., systemic scleroderma, other digestive malabsorption syndromes, and insulin dependent diabetes) No other primary or recurrent invasive cancer within the past 10 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy Endocrine therapy: No concurrent estrogen replacement therapy, including vaginal estrogen creams Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No concurrent enrollment in another clinical trial that has dietary restrictions or endpoints similar to this study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who were diagnosed with early-stage breast cancer within the previous 4 years, and are between the ages of 18-74
Sampling Method: Non-Probability Sample
Enrollment: 3088 (Actual)
Dates: Start 1995-03; Primary Completion 2007-03 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Recurrence | Lifetime

SECONDARY OUTCOMES:
Mortality | Lifetime

CONTACTS AND LOCATIONS:
Overall Officials: John P. Pierce, PhD, Study Chair — University of California, San Diego
Locations (7):
- United States (7):
  - Arizona Cancer Center, Tucson, Arizona
  - University of California San Diego Cancer Center, La Jolla, California
  - Permanente Medical Group (060), Oakland, California
  - University of California Davis School of Medicine, Sacramento, California
  - Northern California Cancer Center, Union City, California
  - Center for Health Research - Portland, Portland, Oregon
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Hyder JA, Thomson CA, Natarajan L, Madlensky L, Pu M, Emond J, Kealey S, Rock CL, Flatt SW, Pierce JP; WHEL Study Group. Adopting a plant-based diet minimally increased food costs in WHEL Study. Am J Health Behav. 2009 Sep-Oct;33(5):530-9. doi: 10.5993/ajhb.33.5.6. PMID 19296743
- [Background] Yost KJ, Haan MN, Levine RA, Gold EB. Comparing SF-36 scores across three groups of women with different health profiles. Qual Life Res. 2005 Jun;14(5):1251-61. doi: 10.1007/s11136-004-6673-8. PMID 16047501
- [Result] Caan BJ, Emond JA, Su HI, Patterson RE, Flatt SW, Gold EB, Newman VA, Rock CL, Thomson CA, Pierce JP. Effect of postdiagnosis weight change on hot flash status among early-stage breast cancer survivors. J Clin Oncol. 2012 May 1;30(13):1492-7. doi: 10.1200/JCO.2011.36.8597. Epub 2012 Mar 19. PMID 22430275
- [Result] Nechuta SJ, Caan BJ, Chen WY, Lu W, Chen Z, Kwan ML, Flatt SW, Zheng Y, Zheng W, Pierce JP, Shu XO. Soy food intake after diagnosis of breast cancer and survival: an in-depth analysis of combined evidence from cohort studies of US and Chinese women. Am J Clin Nutr. 2012 Jul;96(1):123-32. doi: 10.3945/ajcn.112.035972. Epub 2012 May 30. PMID 22648714
- [Result] Al-Delaimy WK, Flatt SW, Natarajan L, Laughlin GA, Rock CL, Gold EB, Caan BJ, Parker BA, Pierce JP. IGF1 and risk of additional breast cancer in the WHEL study. Endocr Relat Cancer. 2011 Mar 3;18(2):235-44. doi: 10.1530/ERC-10-0121. Print 2011 Apr. PMID 21263044
- [Result] Bertram LA, Stefanick ML, Saquib N, Natarajan L, Patterson RE, Bardwell W, Flatt SW, Newman VA, Rock CL, Thomson CA, Pierce JP. Physical activity, additional breast cancer events, and mortality among early-stage breast cancer survivors: findings from the WHEL Study. Cancer Causes Control. 2011 Mar;22(3):427-35. doi: 10.1007/s10552-010-9714-3. Epub 2010 Dec 24. PMID 21184262
- [Result] Emond JA, Patterson RE, Natarajan L, Laughlin GA, Gold EB, Pierce JP. Sex hormone concentrations and the risk of breast cancer recurrence in postmenopausal women without hot flashes. Cancer Epidemiol Biomarkers Prev. 2011 May;20(5):939-45. doi: 10.1158/1055-9965.EPI-10-1240. Epub 2011 Mar 17. PMID 21415358
- [Result] Jacobs ET, Thomson CA, Flatt SW, Al-Delaimy WK, Hibler EA, Jones LA, Leroy EC, Newman VA, Parker BA, Rock CL, Pierce JP. Vitamin D and breast cancer recurrence in the Women's Healthy Eating and Living (WHEL) Study. Am J Clin Nutr. 2011 Jan;93(1):108-17. doi: 10.3945/ajcn.2010.30009. Epub 2010 Oct 27. PMID 20980485
- [Result] Madlensky L, Natarajan L, Tchu S, Pu M, Mortimer J, Flatt SW, Nikoloff DM, Hillman G, Fontecha MR, Lawrence HJ, Parker BA, Wu AH, Pierce JP. Tamoxifen metabolite concentrations, CYP2D6 genotype, and breast cancer outcomes. Clin Pharmacol Ther. 2011 May;89(5):718-25. doi: 10.1038/clpt.2011.32. Epub 2011 Mar 23. PMID 21430657
- [Result] Paxton RJ, Jones LA, Chang S, Hernandez M, Hajek RA, Flatt SW, Natarajan L, Pierce JP. Was race a factor in the outcomes of the Women's Health Eating and Living Study? Cancer. 2011 Aug 15;117(16):3805-13. doi: 10.1002/cncr.25957. Epub 2011 Feb 11. PMID 21319157
- [Result] Gold EB, Pierce JP, Natarajan L, Stefanick ML, Laughlin GA, Caan BJ, Flatt SW, Emond JA, Saquib N, Madlensky L, Kealey S, Wasserman L, Thomson CA, Rock CL, Parker BA, Karanja N, Jones V, Hajek RA, Pu M, Mortimer JE. Dietary pattern influences breast cancer prognosis in women without hot flashes: the women's healthy eating and living trial. J Clin Oncol. 2009 Jan 20;27(3):352-9. doi: 10.1200/JCO.2008.16.1067. Epub 2008 Dec 15. PMID 19075284
- [Result] Pierce JP, Natarajan L, Caan BJ, Flatt SW, Kealey S, Gold EB, Hajek RA, Newman VA, Rock CL, Pu M, Saquib N, Stefanick ML, Thomson CA, Parker B. Dietary change and reduced breast cancer events among women without hot flashes after treatment of early-stage breast cancer: subgroup analysis of the Women's Healthy Eating and Living Study. Am J Clin Nutr. 2009 May;89(5):1565S-1571S. doi: 10.3945/ajcn.2009.26736F. Epub 2009 Apr 1. PMID 19339393
- [Result] Rock CL, Natarajan L, Pu M, Thomson CA, Flatt SW, Caan BJ, Gold EB, Al-Delaimy WK, Newman VA, Hajek RA, Stefanick ML, Pierce JP; Women's Healthy Eating and Living Study Group. Longitudinal biological exposure to carotenoids is associated with breast cancer-free survival in the Women's Healthy Eating and Living Study. Cancer Epidemiol Biomarkers Prev. 2009 Feb;18(2):486-94. doi: 10.1158/1055-9965.EPI-08-0809. Epub 2009 Feb 3. PMID 19190138
- [Result] Hernandez-Valero MA, Thomson CA, Hernandez M, Tran T, Detry MA, Theriault RL, Hajek RA, Pierce JP, Flatt SW, Caan BJ, Jones LA. Comparison of baseline dietary intake of Hispanic and matched non-Hispanic white breast cancer survivors enrolled in the Women's Healthy Eating and Living study. J Am Diet Assoc. 2008 Aug;108(8):1323-9. doi: 10.1016/j.jada.2008.05.008. PMID 18656572
- [Result] Mortimer JE, Flatt SW, Parker BA, Gold EB, Wasserman L, Natarajan L, Pierce JP; WHEL Study Group. Tamoxifen, hot flashes and recurrence in breast cancer. Breast Cancer Res Treat. 2008 Apr;108(3):421-6. doi: 10.1007/s10549-007-9612-x. Epub 2007 May 31. PMID 17541741
- [Result] Saxe GA, Madlensky L, Kealey S, Wu DP, Freeman KL, Pierce JP. Disclosure to physicians of CAM use by breast cancer patients: findings from the Women's Healthy Eating and Living Study. Integr Cancer Ther. 2008 Sep;7(3):122-9. doi: 10.1177/1534735408323081. PMID 18956493
- [Result] Hong S, Bardwell WA, Natarajan L, Flatt SW, Rock CL, Newman VA, Madlensky L, Mills PJ, Dimsdale JE, Thomson CA, Hajek RA, Chilton JA, Pierce JP. Correlates of physical activity level in breast cancer survivors participating in the Women's Healthy Eating and Living (WHEL) Study. Breast Cancer Res Treat. 2007 Jan;101(2):225-32. doi: 10.1007/s10549-006-9284-y. Epub 2006 Sep 21. PMID 17028988
- [Result] Parker BA, Flatt SW, Mortimer JA, et al.: Impact of hormone replacement therapy on breast cancer: Women's Healthy Eating and Living (WHEL) study experience. [Abstract] Breast Cancer Res Treat 106 (1): A-1055, S59, 2007.
- [Result] Pierce JP, Natarajan L, Caan BJ, Parker BA, Greenberg ER, Flatt SW, Rock CL, Kealey S, Al-Delaimy WK, Bardwell WA, Carlson RW, Emond JA, Faerber S, Gold EB, Hajek RA, Hollenbach K, Jones LA, Karanja N, Madlensky L, Marshall J, Newman VA, Ritenbaugh C, Thomson CA, Wasserman L, Stefanick ML. Influence of a diet very high in vegetables, fruit, and fiber and low in fat on prognosis following treatment for breast cancer: the Women's Healthy Eating and Living (WHEL) randomized trial. JAMA. 2007 Jul 18;298(3):289-98. doi: 10.1001/jama.298.3.289. PMID 17635889
- [Result] Pierce JP, Natarajan L, Cann BJ, et al.: The influence of a very high vegetable-fruit-fiber, low-fat diet on prognosis following treatment for breast cancer: results from the Womens Healthy Eating and Living (WHEL) randomized trial. [Abstract] Breast Cancer Res Treat 106 (1): A-61, S16, 2007.
- [Result] Pierce JP, Stefanick ML, Flatt SW, Natarajan L, Sternfeld B, Madlensky L, Al-Delaimy WK, Thomson CA, Kealey S, Hajek R, Parker BA, Newman VA, Caan B, Rock CL. Greater survival after breast cancer in physically active women with high vegetable-fruit intake regardless of obesity. J Clin Oncol. 2007 Jun 10;25(17):2345-51. doi: 10.1200/JCO.2006.08.6819. PMID 17557947
- [Result] Saquib N, Flatt SW, Natarajan L, Thomson CA, Bardwell WA, Caan B, Rock CL, Pierce JP. Weight gain and recovery of pre-cancer weight after breast cancer treatments: evidence from the women's healthy eating and living (WHEL) study. Breast Cancer Res Treat. 2007 Oct;105(2):177-86. doi: 10.1007/s10549-006-9442-2. Epub 2006 Nov 23. PMID 17123151
- [Result] Bardwell WA, Natarajan L, Dimsdale JE, Rock CL, Mortimer JE, Hollenbach K, Pierce JP. Objective cancer-related variables are not associated with depressive symptoms in women treated for early-stage breast cancer. J Clin Oncol. 2006 Jun 1;24(16):2420-7. doi: 10.1200/JCO.2005.02.0081. Epub 2006 May 1. PMID 16651649
- [Result] Madlensky L, Flatt SW, Bardwell WA, Rock CL, Pierce JP; WHEL Study group. Is family history related to preventive health behaviors and medical management in breast cancer patients? Breast Cancer Res Treat. 2005 Mar;90(1):47-54. doi: 10.1007/s10549-004-2626-8. PMID 15770526
- [Result] Newman VA, Thomson CA, Rock CL, Flatt SW, Kealey S, Bardwell WA, Caan BJ, Pierce JP; Women's Healthy Eating and Living (WHEL) Study Group. Achieving substantial changes in eating behavior among women previously treated for breast cancer--an overview of the intervention. J Am Diet Assoc. 2005 Mar;105(3):382-91; quiz 488. doi: 10.1016/j.jada.2004.12.008. PMID 15746825
- [Result] Thomson CA, Giuliano AR, Shaw JW, Rock CL, Ritenbaugh CK, Hakim IA, Hollenbach KA, Alberts DS, Pierce JP. Diet and biomarkers of oxidative damage in women previously treated for breast cancer. Nutr Cancer. 2005;51(2):146-54. doi: 10.1207/s15327914nc5102_4. PMID 15860436
- [Result] Thornton AA, Madlensky L, Flatt SW, Kaplan RM, Pierce JP. The impact of a second breast cancer diagnosis on health related quality of life. Breast Cancer Res Treat. 2005 Jul;92(1):25-33. doi: 10.1007/s10549-005-1411-7. PMID 15980988
- [Result] Pierce JP, Newman VA, Flatt SW, Faerber S, Rock CL, Natarajan L, Caan BJ, Gold EB, Hollenbach KA, Wasserman L, Jones L, Ritenbaugh C, Stefanick ML, Thomson CA, Kealey S; Women's Healthy Eating and Living (WHEL) Study Group. Telephone counseling intervention increases intakes of micronutrient- and phytochemical-rich vegetables, fruit and fiber in breast cancer survivors. J Nutr. 2004 Feb;134(2):452-8. doi: 10.1093/jn/134.2.452. PMID 14747688
- [Result] Rock CL, Flatt SW, Thomson CA, Stefanick ML, Newman VA, Jones L, Natarajan L, Pierce JP, Chang RJ, Witztum JL; Women's Healthy Eating and Living (WHEL) Study Group. Plasma triacylglycerol and HDL cholesterol concentrations confirm self-reported changes in carbohydrate and fat intakes in women in a diet intervention trial. J Nutr. 2004 Feb;134(2):342-7. doi: 10.1093/jn/134.2.342. PMID 14747670
- [Result] Gold EB, Flatt SW, Pierce JP, Bardwell WA, Hajek RA, Newman VA, Rock CL, Stefanick ML. Dietary factors and vasomotor symptoms in breast cancer survivors: the WHEL Study. Menopause. 2006 May-Jun;13(3):423-33. doi: 10.1097/01.gme.0000185754.85328.44. PMID 16735939
- [Result] Pierce JP, Faerber S, Wright FA, Rock CL, Newman V, Flatt SW, Kealey S, Jones VE, Caan BJ, Gold EB, Haan M, Hollenbach KA, Jones L, Marshall JR, Ritenbaugh C, Stefanick ML, Thomson C, Wasserman L, Natarajan L, Thomas RG, Gilpin EA; Women's Healthy Eating and Living (WHEL) study group. A randomized trial of the effect of a plant-based dietary pattern on additional breast cancer events and survival: the Women's Healthy Eating and Living (WHEL) Study. Control Clin Trials. 2002 Dec;23(6):728-56. doi: 10.1016/s0197-2456(02)00241-6. PMID 12505249
- [Result] Wasserman L, Flatt SW, Natarajan L, Laughlin G, Matusalem M, Faerber S, Rock CL, Barrett-Connor E, Pierce JP. Correlates of obesity in postmenopausal women with breast cancer: comparison of genetic, demographic, disease-related, life history and dietary factors. Int J Obes Relat Metab Disord. 2004 Jan;28(1):49-56. doi: 10.1038/sj.ijo.0802481. PMID 14557830